CLINICAL TRIAL: NCT00140478
Title: A Phase II Study of Mifepristone (RU-486) in Androgen Independent Prostate Cancer With Correlative Assessment of Androgen Receptor Co-Repressor Proteins
Brief Title: Mifepristone (RU-486) in Androgen Independent Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Massachusetts General Hospital (Other); Brigham and Women's Hospital (Other); Georgetown University (Other)
Responsible Party: Mary-Ellen Taplin, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-249
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2009-12-09 (Estimated); Status verified 2009-12

CONDITIONS: Prostate Cancer; Adenocarcinoma of Prostate
Keywords: Androgen Independent Prostate Cancer; Prostate Cancer; Mifepristone; RU-486
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Mifepristone

INTERVENTIONS:
Drug: Mifepristone — 200mg orally once daily
  Other Names: RU-486

SUMMARY:
The purpose of this study is to determine the effects (good and bad) that mifepristone has on patients with androgen independent prostate cancer.

DETAILED DESCRIPTION:
Patients will receive mifepristone, 200mg orally once a day. One treatment cycle is 28 days long. Patients will remain on treatment unless their cancer gets worse or they develop intolerable side effects.

At the end of each cycle a physical examination, routine blood tests, and hormone levels will be performed.

After every 3 cycles, one or more of the following will be performed: bone scan, chest x-ray, CT scan or MRI.

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation of adenocarcinoma of the prostate
* Bone metastasis(es) by bone scan or cat scan
* Clinical, biochemical, or radiographic progression after primary androgen ablation with either orchiectomy or gonadotropin releasing hormone analog therapy.
* One prior chemotherapy treatment is allowed.
* > 3 weeks since major surgery
* > 4 weeks since radiotherapy
* > 8 weeks since prior strontium-89 or samarium 153
* ECOG performance status 0 or 1
* Absolute neutrophil count (ANC) > 1,500/ul
* Platelets > 100,000/ul
* Bilirubin < 1.5 x upper limit of normal (ULN)
* AST or ALT < 3 x ULN
* Creatinine < 1.5 x ULN
* Electrolytes within 10% of normal range
* Serum testosterone < 50ng/dL
* Prostate-specific antigen (PSA) > 5.0ng/ml

Exclusion Criteria:

* Concomitant therapy with corticosteroids
* Chemotherapy within 28 days
* Currently active second malignancy other than non-melanoma skin cancer
* Baseline adrenal insufficiency requiring long-term steroids

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2005-02; Primary Completion 2006-06 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
To determine the therapeutic efficacy of mifepristone in patients with androgen independent prostate cancer | 2 years

SECONDARY OUTCOMES:
To determine the duration of response, time to disease progression and safety of mifepristone in patients with androgen independent prostate cancer

CONTACTS AND LOCATIONS:
Overall Officials: Mary-Ellen Taplin, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Georgetown University, Washington D.C., District of Columbia
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts